CLINICAL TRIAL: NCT04219150
Title: Comparative Study Between Cardiometry Versus Fluid and Catheter Treatment Trial (FACTT Lite) on Fluid Management in Acute Respiratory Distress Syndrome Patients
Brief Title: Cardiometry Versus Fluid and Catheter Treatment Trial (FACTT Lite) on Fluid Management in Acute Respiratory Distress Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Shaheen, Assistant lecturer of Anesthesiology, Surgical ICU and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32721/11/18
Record Dates: First submitted 2019-12-22; First posted 2020-01-06 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: ARDS; Fluid Management; Cardiometry
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical cardiometry (EC) (Experimental)
  Interventions: Device: Electrical cardiometry
- Fluid and Catheter Treatment Trial "FACTT Lite" (Experimental)
  Interventions: Drug: Fluid and Catheter Treatment Trial "FACTT Lite"

INTERVENTIONS:
Device: Electrical cardiometry — Four sensors of EC will be applied : first approximately 5 cm above the base of the neck, second on the base of neck, third on the lower thorax at the level of the xiphoid and the fourth one on the lower thorax approximately 5 cm below the 3rd electrode at the level of anterior axillary line. The EC monitor (Electrical Cardiometry monitor, ICON Cardiotronics, Inc., La Jolla, CA 92307; Osyka Medical GmbH, Berlin, and Germany, model C3, serial number 1725303) will be connected to the sensor cable and the patient data will be fed. Corrected flow time (FTC) and stroke volume (SV) will be measured continuously in less than 30 seconds after placing the sensors and inputting the height and weight.
  Arms: Electrical cardiometry (EC)
Drug: Fluid and Catheter Treatment Trial "FACTT Lite" — The FACTT Lite provided three possible instructions determined by the CVP and urine output: furosemide administration, fluid bolus, or no intervention. FACTT Lite contained instructions to withhold furosemide until the patient achieved a mean arterial pressure greater than 60 mmHg off of vasopressors for at least 12 h.
  Arms: Fluid and Catheter Treatment Trial "FACTT Lite"

SUMMARY:
The aim of this study will be to compare the fluid management in acute respiratory distress syndrome ARDS guided by electrical cardiometry (EC) versus the guidance with simplified conservative fluid protocol, Fluid and Catheter Treatment Trial "FACTT Lite". Group (A) consists of 35 patients: Fluid management in this group will follow a simplified conservative fluid protocol, "FACTT Lite" The FACTT Lite provided three possible instructions determined by the CVP and urine output: furosemide administration, fluid bolus, or no intervention. Group (B) consists of 35 patients: Fluid will be allowed according to an FTc-based fluids algorithm protocol and the type of bolus fluids will be determined according to Transthoracic fluid content (TFC), vasopressors and inotropes will be given according to reading of EC reading of systemic vascular resistance (SVR) and index of contractility (I CON).

ELIGIBILITY:
Inclusion Criteria:

* Acute onset within one week
* Mild to moderate ARDS (FiO2/PaO2) less than 300 mmHg and more than 100 mmHg with a minimum PEEP of 5 cmH2O
* Bilateral lung opacities consistent with pulmonary edema on chest radiogram or lung ultrasound, cardiac failure, and fluid overload should be excluded in the absence of a definite cause of ARDS
* ARDS due to pulmonary cause.

Exclusion Criteria:

* Hemodynamic instability, patients on vasopressor,
* Barotrauma
* organ/s dysfunction at presentation.
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Percentage of mortality at 28th day | 28 day
  Percentage of mortality at 28th day in each group

SECONDARY OUTCOMES:
Oxygenation index | 28 day
  Higher scores mean a better outcome.
Lung injury score | 28 day
  Higher scores mean a worse outcome.
Duration of mechanical ventilation | 28 day
  Duration of mechanical ventilation (days) in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol